CLINICAL TRIAL: NCT04655339
Title: Efficacy of Laparoscopic Transversus Abdominis Plane (TAP) Block to Reduce Post-operative Opioids Following Bariatric and Minimally Invasive Foregut Surgery
Brief Title: Laparoscopic Transversus Abdominis Plane (TAP) Block to Reduce Post-operative Opioids
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was not started due to COVID-19 pandemic.
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 019-428
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group-1 (Experimental): Bilateral abdominal Lap-TAP block injection near incision site with 0.25% Bupivacaine HCl (30cc) with 30ml being injected bilaterally. Remaining residual is injected into port incision sites.
  Interventions: Drug: Bilateral abdominal Lap-TAP
- Group-2 (Experimental): Bilateral abdominal Lap-TAP liposomal Bupivacaine (Exparel®) injection with 133mg (20ml) Exparel® plus bupivacaine 0.25% (30ml), plus 10ml of normal saline for a total volume of 60ml, injecting 30ml each side.
  Interventions: Drug: Bilateral abdominal Lap-TAP
- Group-3 (No Intervention): No intervention

INTERVENTIONS:
Drug: Bilateral abdominal Lap-TAP — Subjects will have Liposomal Bupivacaine (Exparel®) or the control injected into the transversus abdominis plane bilaterally.
  Arms: Group-1; Group-2

SUMMARY:
This study evaluates laparoscopic-guided TAP block for reducing opioid use after minimally invasive foregut and bariatric surgeries, comparing Bupivacaine HCL with Exparel®. Secondary outcomes include pain scores, length of stay, and PONV medication use.

DETAILED DESCRIPTION:
In this study the investigators aim to investigate the efficacy of laparoscopic-guided TAP block in reducing post-operative opioid use following minimally invasive foregut and bariatric surgeries. The investigators will also compare and report the analgesia produced by Bupivacaine HCL vs Exparel ®, a prolonged slow release Liposomal Bupivacaine formulation. Secondary outcomes assessed will be VAS pain scores, length of stay, and PONV dosage administered.

ELIGIBILITY:
Inclusion Criteria:

* gastric bypass & sleeve gastrectomy, duodenal switch and minimally invasive elective anti-reflux foregut surgeries such as - hiatal hernia repair, fundoplication and Heller myotomy.

Exclusion Criteria:

* Subjects who are known to be
* Allergic to Bupivacaine
* Chronic opioid users Page 4
* Had/have neurological conditions
* Have a diagnosis of chronic pain syndrome which requires them to consume regular analgesics > 3-months
* American Society of Anesthesiologists (ASA) Class IV & V patients with severe systemic disease that is a constant threat to life.
* Patients with abdominal drain use
* Patients with significant cardiovascular, liver or renal disease
* Presence of contraindications for bariatric or foregut surgery.
* Patients presenting postoperative complications will be excluded from final analysis & final data set
* History of bariatric or foregut surgery
* Patients who are pregnant
* Patients who are under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
opioid dosage requested | 30days
  opioid dosage requested post-TAP block

SECONDARY OUTCOMES:
visual analog scores (VAS) | 30days
length of stay | 30days
anti-emetic dosage | 30days

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No